CLINICAL TRIAL: NCT05741502
Title: An Exploratory Analysis of Immune and Inflammatory Response Associated with Clozapine Versus Non-Clozapine Antipsychotics in Individuals with Treatment-resistant Schizophrenia
Brief Title: An Exploratory Analysis of Immune and Inflammatory Response Associated with Clozapine
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Walter Stearns, Assistant Clinical Professor, Ohio State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021H0388
Record Dates: First submitted 2023-01-20; First posted 2023-02-23 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Treatment-resistant Schizophrenia
MeSH Terms: conditions — Schizophrenia, Treatment-Resistant | interventions — Clozapine; Antipsychotic Agents; Risperidone; Paliperidone Palmitate; Quetiapine Fumarate; Aripiprazole; ziprasidone; Lurasidone Hydrochloride; cariprazine

STUDY DESIGN:
Intervention Model Description: Parallel open-label groups of Treatment-Refractory schizophrenia patients treated with Clozapine or non-Clozapine drug
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Clozapine Arm (Experimental): Patients will be on Clozapine for at least 6 months
  Interventions: Drug: Clozapine
- Non-Clozapine arm (Active Comparator): Patients will be on non-Clozapine antipsychotic for at least 6 months
  Interventions: Drug: Antipsychotics,Other (non-Clozapine)

INTERVENTIONS:
Drug: Clozapine — We will assess inflammatory/immune marker labs
  Arms: Clozapine Arm
Drug: Antipsychotics,Other (non-Clozapine) — We will assess monitor inflammatory/immune marker lab
  Other Names: Including Olanzapine, Risperidone, Paliperidone, Quetiapine, Aripiprazole, Ziprasidone, Lurasidone, Cariprazine, and all Typical antipsychotics
  Arms: Non-Clozapine arm

SUMMARY:
The specific aim of this protocol is to compare Clozapine treatment vs Non-Clozapine antipsychotic treatment in a population of treatment-refractory individuals with schizophrenia. Specifically, it is to test if Clozapine leads to a decrease in levels of inflammatory markers, namely interleukin-6 but with an exploratory view of other markers. Clozapine has superior efficacy and is the only medication approved for treatment-refractory schizophrenia in addition to decreasing the risk of suicidal behavior as well. It is unclear why Clozapine has increased efficacy from a mechanistic viewpoint. We will look at the role of inflammatory markers and assess them 1x along with rating scales for psychosis and suicidality, the other entities which Clozapine has been shown to improve.

DETAILED DESCRIPTION:
This study is designed to investigate if treatment with the antipsychotic Clozapine is associated with changes in various immune and inflammatory biomarkers when compared to treatment with non-Clozapine antipsychotic treatments. Clozapine is a uniquely efficacious treatment of psychotic disorders, the only effective agent in approximately 30-40% of individuals with treatment refractory symptoms. Clozapine, unlike other antipsychotic drugs, often precipitates a unique, multi-systemic inflammatory response most widely recognized in the cardiovascular system but also likely the central nervous system (CNS) which is tied into its unique side effect profile but might also account for its increased efficacy. Schizophrenia spectrum disorders affect about 1% of the population with around 30-40% of those diagnosed with symptoms refractory to standard, non-Clozapine antipsychotic treatment. We will measure various inflammatory markers 1x for patients who are stable outpatients. Participants will be patients with treatment-resistant schizophrenia on clozapine treatment for at least 6 months referred from OSU's outpatient clinic with a comparator group also referred from Ohio State University, having shown treatment resistant symptoms but with provider/patient electing not to use clozapine for clinically relevant reasons and have been on antipsychotic medication for at least 6 months. The study includes 1 visit including symptom rating scale assessments and laboratory draw for collection of serum samples and the visit also having more diagnostic assessments to assure proper enrollment. If the study results are positive meaning there is a difference between the two groups, it would help elucidate the potential mechanisms by which Clozapine works and demonstrates increased efficacy for those with treatment-refractory schizophrenia, a severely debilitating, life long illness with marked disability. This would also allow for further studies to explore this mechanism and the role of inflammation and the immune system as well.

ELIGIBILITY:
Inclusion Criteria:

* All participants:

  * Between 18 and 65 years of age
  * Physically healthy (no clinically significant unstable medical condition as confirmed by medical history and physical examination)
  * Able to give informed consent
  * Treatment-Refractory Schizophrenia

Clozapine treatment group (n = 30) Individuals treated with Clozapine consistently for a minimum of 6 months

Non-Clozapine treatment group Continued treatment with non-Clozapine antipsychotic but would be eligible for Clozapine with the provider/patient electing to not pursue such for clinical reasons, consistently treated for at least 6 months

Exclusion Criteria:

* Clinically significant medical condition; cardiovascular, pulmonary, endocrine, or renal condition requiring in depth medical treatment
* Active or recent (within 4 weeks) bacterial or viral infection
* Chronic viral infection (hepatitis, HIV)
* History of autoimmune, or chronic inflammatory condition
* Current treatment with lithium
* Treatment with Clozapine in the past 6 months
* Current treatment with immunomodulatory or anti-inflammatory therapy
* Vaccination within the past 3 months
* Current alcohol or substance use disorder of moderate or severe severity
* Intellectual disability (i.e. intelligence quotient <70)
* Unwilling or unable to sign informed consent document
* Pregnancy
* Any patient deemed ineligible by PI discretion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-16 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Interleukin-6 (IL-6) | Up to 1 year
  Comparison in interleukin-6 between Clozapine and non-Clozapine group

SECONDARY OUTCOMES:
Other immune/cardiac markers | Up to 1 year
  Comparison in hsCRP, interleukin-1β, interferon-γ, transforming growth factor-β, tumor necrosis factor between Clozapine and non-Clozapine group
Positive and Negative Syndrome symptom Scale | Up to 1 year
  Comparison in psychosis rating scales (PANSS) between Clozapine and non-Clozapine group. Higher scores indicate more severe symptoms of psychosis. Score from 30-210
Self-injurious Thoughts and Behaviors Interviews | Up to 1 year
  Comparison between Clozapine and non-Clozapine group in Suicidality rating scales. Scores on rating will be binary (yes/no) for suicidal ideation and also suicide attempts.

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio State University Harding Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No